CLINICAL TRIAL: NCT01027611
Title: Patient Assessment of Topical Anesthetic Effectiveness for Intravitreal Injections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Illinois Retina Associates (Other)
Responsible Party: John S. Pollack, M.D., Illinois Retina Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jsp-001
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-12

CONDITIONS: Pain
Keywords: Effectiveness of topical pain medicine for control of pain associated with intravitreal injections; Eye discomfort
MeSH Terms: conditions — Pain | interventions — proxymetacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- proparacaine HCL 0.5% (Experimental)
  Interventions: Drug: proparacaine HCL 0.5%
- proparacaine + lidocaine (Experimental)
  Interventions: Drug: proparacaine HCL 0.5% + 4% lidocaine solution
- lidocaine gel (Experimental)
  Interventions: Drug: 3.5% viscous lidocaine gel

INTERVENTIONS:
Drug: proparacaine HCL 0.5%
  Arms: proparacaine HCL 0.5%
Drug: proparacaine HCL 0.5% + 4% lidocaine solution
  Arms: proparacaine + lidocaine
Drug: 3.5% viscous lidocaine gel
  Arms: lidocaine gel

SUMMARY:
There are currently several different commercially available topical eye drops and gels used to reduce eye discomfort (topical anesthetics) during and after eye injections. Dr. Pollack is performing a research study to evaluate three commercially available topical anesthetics (eye numbing treatments) to determine if individuals have a preference for one over the other. The three topical anesthetics being studied are 1) 0.5% proparacaine hydrochloride (generic, Akorn, Inc), 2) 0.5% proparacaine hydrochloride (generic, Akorn, Inc) PLUS 4% lidocaine hydrochloride topical solution (generic, Roxane Laboratories), and 3) 3.5% lidocaine hydrochloride ophthalmic gel (Akten, Akorn, Inc). These eye anesthetics are NOT experimental medications. They are all commercially available topical anesthetics currently used in our offices and their use is widespread among retina specialists throughout the United States. Dr. Pollack will randomly select one topical anesthetic to use and he will ask you to grade your level of pain associated with the injection procedure. Answering these questions should take less than one minute of your time and your identity will NOT be revealed with the results of this study. The results of this study will be used to inform doctors which eye anesthetics patients find most effective for pain control during eye injections.

DETAILED DESCRIPTION:
In this prospective study, 120 sequential patients undergoing 30 and 33 Gauge intravitreal injections were randomly assigned to receive either: proparacaine HCL 0.5% (Group 1), proparacaine HCL 0.5% + 4% lidocaine liquid drops (Group 2); or 3.5% lidocaine gel (Group 3) as topical anesthetic prior to injection. All procedures utilized a lid speculum and 5% povidone iodine. Approximately 10 seconds after injection, patients graded pain associated with the lid speculum, the needle, and with burning sensation on a pain scale of 0 to 10, with 0 representing no pain and 10 representing the patient's worst imaginable pain. They also graded their overall injection procedure experience as Excellent, Very Good, Fair, Poor, or Awful.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intravitreal injection for treatment of eye disease

Exclusion Criteria:

* Eye infection
* Retinal detachment
* Age less than 18 years
* Pregnant
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Injection experience "grade" | Outcome data is obtained approximately 10 seconds after conclusion of procedure

SECONDARY OUTCOMES:
Pain grades for lid speculum, needle insertion, povidone iodine burning/stinging | Outcome data is obtained approximately 10 seconds after conclusion of procedure

CONTACTS AND LOCATIONS:
Overall Officials: John S. Pollack, MD, Study Chair — Illinois Retina Associates
Locations (1):
- Illinois Retina Associates, Joliet, Illinois, United States